CLINICAL TRIAL: NCT03847961
Title: Efficacy and Safety Study of CA330 Hemoadsorption Device on IL-6 Removal in Septic Patients: A Multicenter Randomized Controlled Trial
Brief Title: Efficacy and Safety Study of CA330 Hemoadsorption Device on IL-6 Removal in Septic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Guangzhou First People's Hospital (Other); Zhujiang Hospital (Other); Beijing Chao Yang Hospital (Other); Peking University Shenzhen Hospital (Other); Fujian Provincial Hospital (Other); Wuhan University (Other)
Responsible Party: Principal Investigator, Guan XiangDong, Chief of the Department of Critical Care Medicine, Chairman of the Chinese Society of Critical Care Medicine, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-030-02
Record Dates: First submitted 2019-02-13; First posted 2019-02-20 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Sepsis
Keywords: sepsis; IL-6; hemoperfusion
MeSH Terms: conditions — Sepsis | interventions — Hemoperfusion

STUDY DESIGN:
Intervention Model Description: Eligible patients are stratified by site and randomly assigned in a 1:1 ratio to either CA330 hemoperfusion plus conventional medical therapy group or conventional medical therapy group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group receive routine treatment of sepsis only. All sites agree, when feasible, to follow the tenets of the Surviving Sepsis Campaign clinical practice guidelines for management of sepsis.
- Experimental Group (Experimental): The experimental group receive routine treatment of sepsis combined with hemoperfusion with cytokine adsorption column (CA330).
  Interventions: Device: hemoperfusion with cytokine adsorption column (CA330)

INTERVENTIONS:
Device: hemoperfusion with cytokine adsorption column (CA330) — Hemoperfusion treatments are performed using a perfusion machine via centrally inserted standard dialysis catheters at a prescribed blood flow rate of 100-300ml/min. In the beginning, lower flow rate is recommended, if there is no discomfort, then gradually increases. Each patient received 2 hemoperfusion treatments within 24 hours with a target duration for each treatment of 120-180 minutes (minimum of 120 minutes). The shorter the interval between the two hemoperfusion is, the better. It is suggested that the second hemoperfusion be performed within 0-5 hours after the first one.
  Arms: Experimental Group

SUMMARY:
Sepsis persists to be the leading causes of morbidity and mortality worldwide. Moreover, the magnitude of health care resources utilized when managing septic patients is huge. All these hard facts call for constant efforts to optimize therapy. At present, the definitive therapy is adequate antibiotics and infectious source control. Fortunately, research has led to a better understanding of the pathophysiology of sepsis, in which the activation of multiple pro- and anti-inflammatory mediators plays a key role. This has led to the development of treatment strategies aimed at restoring a balanced immune response by eliminating/deactivating these inflammatory mediators. Whilst animal models of sepsis have provided encouraging results with strategies aiming at immune response modulation, clinical studies in patients using targeted pharmacological approaches have so far proved disappointing.

Besides of acute kidney injury (AKI), renal replacement therapy (RRT) is applied to remove inflammatory mediators extracorporeally. Across the different modalities, the application of adsorption may help deactivate and decrease the peak elevation of these mediators in earlier course of sepsis, when levels of endotoxins and cytokines are extremely high. Recently, attempts to improve the outcome of sepsis patients with such devices, ie CytoSorb cytokine hemoadsorption and polymyxin B (Toraymyxin) endotoxin adsorption, have seen a certain renaissance. However, the clinical evidence to date supporting hemoadsorption for removal of endotoxins and/or proinflammatory mediators in sepsis remains incompetent and controversial.

CA330 (Jafron Biomedical Co , Ltd, Zhuhai, China) is a hemoadsorption device containing hemocompatible, porous polymeric beads capable of removing cytokines and other mid-molecular weight toxins from blood by size exclusion and surface adsorption. Compared with HA330, improved resin synthesis technology makes CA330 a better performance in removing cytokines. This trial is the first to evaluate CA330 efficacy of cytokine reduction using the change in plasma interleukin (IL)-6 concentrations over time as a primary outcome. Although the trial was neither designed nor powered to evaluate outcome, we also evaluated organ function parameters as well as 28-day all-cause mortality.

DETAILED DESCRIPTION:
Eligible patients are stratified by site and randomly assigned in a 1:1 ratio to either CA330 hemoperfusion plus conventional medical therapy group or conventional medical therapy group. The randomization is performed by researchers on the central randomization system, provided by the Department of Biostatistics, Southern Medical University. In this study, the center coded random number table is produced by stratified and sectional randomization method. Statistical Analysis System(SAS) 9.4 statistical software is used to generate random coding tables with serial numbers (001-144) according to the number of cases allocated in each center and the proportion of experimental group and control group (1:1). The length of selected sections (block) and random seed number are sealed together as confidential data . The random number table is provided by the statisticians of the Department of Biostatistics, Southern Medical University.

The experimental group receive routine treatment of sepsis combined with cytokine adsorption column (CA330) perfusion, and the control group receive routine treatment of sepsis only.

Hemoperfusion treatments are performed using a perfusion machine via centrally inserted standard dialysis catheters at a prescribed blood flow rate of 100-300ml/min. In the beginning, lower flow rate is recommended, if there is no discomfort, then gradually increases. Each patient received 2 hemoperfusion treatments within 24 hours with a target duration for each treatment of 120-180 minutes (minimum of 120 minutes). The shorter the interval between the two hemoperfusion is, the better. It is suggested that the second hemoperfusion be performed within 0-5 hours after the first one.

Anticoagulation was recommended with low-molecular-weight heparin in arterial line of the circuit at the dose of 60-80 international units (IU)/kg. No additional dose is required. The activity of anticoagulant factor α can be monitored at 60 minutes. It is suggested that the activity of anticoagulant factor α should be maintained at 500-1000units/L in subjects without bleeding tendency and 200-400units/L in subjects with bleeding tendency. If the clinical condition is limited, it is not mandatory to monitor this parameter.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients aged 18-75 years, regardless of gender;
2. Meet the clinical criteria of sepsis according to the Third International Consensus Definitions for Sepsis;
3. The diagnosis of sepsis is established within last 48 hours.
4. Written informed consent is signed, and agreement to participate in all visits, examinations and treatments as required by the research program is achieved. If a patient is not able to give consent, the legal representative is asked to consent.

Exclusion Criteria:

1. End-stage renal disease that need maintenance hemodialysis treatment;
2. Congenital or acquired immunodeficiency disorders or those who had received organ transplantation within one year;
3. Prescription of immunosuppressive medications (tripterygium wilfordii, mycophenolate mofetil, cyclophosphamide, FK506, etc.) or prednisolone for more than 10 mg/day (or the same dose of other hormone therapy) within 30 days;
4. Coagulation dysfunction, severe bleeding tendency (prothrombin time, activated partial thromboplastin time prolonged significantly with bleeding, or fibrinogen less than 1.2 g/L with bleeding), active bleeding or uncontrolled acute massive bleeding within 24 hours;
5. Malignant tumors, consumptive diseases, site of infection cannot be cleared (ie surgical patients who cannot be operated on) or body weight less than 35kg;
6. A terminal state of organ failure (end stage of chronic obstructive pulmonary disease, pulmonary heart disease, heart dysfunction stage-IV, brain death or persistent vegetative state, chronic liver disease with hepatic encephalopathy, coagulation dysfunction, fluid retention and hepatocellular jaundice);
7. Following results are detected during screening: platelet count < 50 *10^9/L, neutrophil count < 0.5 *10^9/L, hemoglobin < 70 g/L;
8. Despite of adequate volume resuscitation, vasopressors and hormones, the mean arterial blood cannot maintain above 65 mmHg;
9. Those who have been participating in or participated in another interventional clinical study within 30 days prior to enrollment, such as the clinical study of related drugs or medical devices affecting immunity (ie Xuebijing, ulinastatin, continuous renal replacement therapy, etc.);
10. Anaphylaxis to materials of cardiopulmonary bypass, anticoagulants and hemoperfusion or other serious allergic history;
11. Those who are not suitable for this clinical trial, which is determined by researchers, such as pregnant or lactating women, current drug addicts, patients with severe mental or neurological disorders, and those who have a history of alcohol abuse and cannot be terminated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
the reduction rate of IL-6 serum concentration at the initiation of first adsorption and at the end of the second adsorption | from the initiation of first adsorption until the end of the second adsorption, assessed up to 24hours
  (1-Concentration IL-6 end of second adsorption/ Concentration IL-6 initiation of first adsorption) ×100%

SECONDARY OUTCOMES:
the reduction rate of IL-10 serum concentration at the initiation of first adsorption and at the end of the second adsorption | from the initiation of first adsorption until the end of the second adsorption, assessed up to 24hours
  (1-Concentration IL-10 end of second adsorption/ Concentration IL-10 initiation of first adsorption) ×100%
the reduction rate of lactic acid serum concentration at the initiation of first adsorption and at the end of the second adsorption | from the initiation of first adsorption until the end of the second adsorption, assessed up to 24hours
  (1-Concentration lactic acid end of second adsorption/ Concentration lactic acid initiation of first adsorption) ×100%
the reduction rate of tumor necrosis factor-α (TNF-α) serum concentration at the initiation of first adsorption and at the end of the second adsorption | from the initiation of first adsorption until the end of the second adsorption, assessed up to 24hours
  (1-Concentration TNF-α end of second adsorption/ Concentration TNF-α initiation of first adsorption) ×100%
the dynamic change of Acute Physiology and Chronic Health Evaluation (APACHE II) score | from Day0 to Day28
  The maximum APACHE II score is 71, while the minimum score is 0. The higher values represent a worse outcome.
ventilation time | from Day0 to Day28
  scale: hour
oxygenation index | from Day0 to Day28
  partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2)
24hour urinary output | from Day0 to Day28
  scale: ml/24h
length of vasopressors | from Day0 to Day28
  scale: hour
catecholamine index | from Day0 to Day28
  (dopamine dose*1)+(dobutamine dose*1)+(adrenaline dose*100)+(noradrenaline dose*100)+(phenylephrine dose*100), wherein all doses are expressed as µg/kg/min.
RRT incidency | from Day0 to Day28
  the percentages of patients who receive RRT in two groups
total length of renal replacement therapy | from Day0 to Day28
  scale: hour
ICU and hospital length of stay | from Day0 to Day28
  scale: day
28-day all-cause mortality | from Day0 to Day28
  the 28-day all-cause mortality in two groups

OTHER OUTCOMES:
body temperature | from Day0 to Day28
  scale: ℃
heart rate | from Day0 to Day28
  scale: beats per minute (bpm)
respiratory rate | from Day0 to Day28
  scale: times per minute
blood pressure | from Day0 to Day28
  Both systolic and diastolic pressure will be measured. Scale: mmHg
count of white blood cell | from Day0 to Day28
  scale: cells/L
count of neutrophils | from Day0 to Day28
  scale: cells/L
concentration of hemoglobin | from Day0 to Day28
  scale: g/dl
hematocrit value | from Day0 to Day28
  hematocrit value
count of platelet | from Day0 to Day28
  scale: cells/L
prothrombin time (PT) | from Day0 to Day28
  scale: second
activated partial thromboplastin time (APPT) | from Day0 to Day28
  scale: second
level of fibrinogen | from Day0 to Day28
  scale: g/dl
thrombin time (TT) | from Day0 to Day28
  scale: second
level of serum Alanine transaminase (ALT) | from Day0 to Day28
  scale: Unit/L (U/L)
level of serum Aspartate transaminase (AST) | from Day0 to Day28
  scale: Unit/L (U/L)
level of total bilirubin | from Day0 to Day28
  scale: µmol/L
level of direct bilirubin | from Day0 to Day28
  scale: µmol/L
level of total protein | from Day0 to Day28
  scale: g/L
level of albumin | from Day0 to Day28
  scale: g/L
concentration of serum creatinine | from Day0 to Day28
  scale: mg/dl
concentration of blood urea nitrogen | from Day0 to Day28
  scale: mmol/L
concentration of serum potassium | from Day0 to Day28
  scale: mmol/L
concentration of serum sodium | from Day0 to Day28
  scale: mmol/L
concentration of serum calcium | from Day0 to Day28
  scale: mmol/L
concentration of serum phosphorus | from Day0 to Day28
  scale: mmol/L
concentration of serum magnesium | from Day0 to Day28
  scale: mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Guan, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China